CLINICAL TRIAL: NCT01427933
Title: An Open-Label, Multicenter, Randomized, Phase 2 Study Evaluating the Efficacy and Safety of Ramucirumab (IMC-1121B) Drug Product in Combination With Eribulin Versus Eribulin Monotherapy in Unresectable, Locally-Recurrent or Metastatic Breast Cancer Patients Previously Treated With Anthracycline and Taxane Therapy
Brief Title: A Study of Ramucirumab (IMC-1121B) in Combination With Eribulin Versus Eribulin Alone in Participants With Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14392; I4T-IE-JVCD (Other: Eli Lilly and Company); CP12-1134 (Other: Imclone Systems)
Record Dates: First submitted 2011-08-31; First posted 2011-09-02 (Estimated); Results first posted 2014-08-19 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2016-12

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Ramucirumab; eribulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ramucirumab and Eribulin (Experimental): Ramucirumab 10 milligrams/kilogram (mg/kg) administered by intravenous (IV) infusion on Day 1 of each 3-week cycle
  Eribulin 1.4 milligrams/square meter (mg/m²) administered by IV bolus on Day 1 and Day 8 of each 3-week cycle
  Interventions: Biological: Ramucirumab (IMC-1121B); Drug: Eribulin
- Eribulin Monotherapy (Active Comparator): Eribulin 1.4 mg/m² administered by IV bolus on Day 1 and Day 8 of each 3-week cycle
  Interventions: Drug: Eribulin

INTERVENTIONS:
Biological: Ramucirumab (IMC-1121B) — Administered intravenously
  Other Names: LY3009806
  Arms: Ramucirumab and Eribulin
Drug: Eribulin — Administered intravenously

SUMMARY:
This is a study to compare the antitumor activity of ramucirumab (IMC-1121B) and eribulin together versus eribulin alone, in participants with locally recurrent or metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Have histologically or cytologically confirmed invasive breast cancer which at the time of study entry is either locally recurrent disease not amenable to curative therapy or Stage IV disease (American Joint Committee on Cancer Staging Criteria for breast cancer)
* Have measurable and/or nonmeasurable disease per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1)
* Have received at least 2 but not more than 4 prior cytotoxic chemotherapy regimens in the locally recurrent or metastatic setting
* Have received prior treatment with both anthracyclines and taxanes, either in the metastatic, adjuvant or neoadjuvant setting
* Have received Human Epidermal Growth Factor Receptor 2 (HER-2) directed treatment; or are not a candidate for HER-2-directed treatment if the patient has HER-2 positive disease
* Have completed any prior radiotherapy and/or hormonal therapy at least 1 week prior to randomization and have recovered from all clinically significant treatment-related toxicities
* Have an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Have left ventricular ejection fraction within normal limits
* Have discontinued all previous chemotherapy treatments for cancer at least 3 weeks prior to randomization and recovered from clinically significant toxic effects
* Have resolution to Grade less than or equal to 1 [by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE), Version 4.0] of all clinically significant toxicities of prior chemotherapy, surgery, radiotherapy, or hormonal therapy with the exception of peripheral neuropathy, which must have resolved to Grade less than or equal to 2
* Have adequate hematologic, hepatic, renal, and coagulation function
* Test negative for pregnancy
* Have a life expectancy of at least 3 months

Exclusion Criteria:

* Have a concurrent active other malignancy other than adequately treated non-melanomatous skin cancer or other noninvasive or in situ neoplasms
* Are currently enrolled in, or recently discontinued from, a clinical trial involving an investigational product, or concurrently enrolled in any other type of medical research judged not to be medically compatible with the study
* Have received investigational therapy within 3 weeks prior to randomization
* Have received prior ramucirumab or eribulin
* Have a known sensitivity to agents of similar biologic composition as ramucirumab, halichondrin B and/or halichondrin B chemical derivative
* Have received bevacizumab within 6 weeks prior to randomization
* Have uncontrolled or poorly controlled hypertension
* Have congenital prolonged QTc syndrome (or have a family history) or prolongation of QTc at baseline
* Have a history of additional risk factors for torsades de pointes within the last year prior to randomization
* Have an implantable pacemaker or automatic implantable cardioverter defibrillator
* Have bradycardia
* Have an acute/subacute bowel obstruction or history of chronic diarrhea requiring ongoing medical intervention within 6 months prior to randomization
* Have a history of uncontrolled hereditary or acquired bleeding or thrombotic disorders
* Have experienced a Grade 3 or greater bleeding event within 3 months prior to randomization
* Have experienced any Grade 3 or greater arterial thromboembolic events within 6 months prior to randomization, or venous thromboembolic event within 3 months prior to randomization
* Have undergone major surgery within 4 weeks prior to randomization or subcutaneous venous access device placement within 7 days prior to randomization
* Have a planned major surgery to be performed during the course of the trial
* Have uncontrolled metabolic conditions
* Have an ongoing or active infection requiring parenteral antibiotic, antifungal, or antiviral therapy
* Have known human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS)
* Have pulmonary lymphangitic involvement that results in pulmonary dysfunction requiring active treatment including the use of oxygen
* Have received a prior allogeneic organ or tissue transplantation
* Have had a serious nonhealing wound, ulcer, or bone fracture within 4 weeks prior to randomization
* Have known leptomeningeal metastases
* Have cirrhosis (Child-Pugh Level B or worse) or cirrhosis (any degree) and a history of hepatic encephalopathy or clinically meaningful ascites

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2011-11; Primary Completion 2013-09 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (52):
- United States (52):
  - ImClone Investigational Site, Birmingham, Alabama
  - ImClone Investigational Site, Gilroy, California
  - ImClone Investigational Site, Palm Springs, California
  - ImClone Investigational Site, Denver, Colorado
  - ImClone Investigational Site, Southington, Connecticut
  - ImClone Investigational Site, Fort Myers, Florida
  - ImClone Investigational Site, Jacksonville, Florida
  - ImClone Investigational Site, Orlando, Florida
  - ImClone Investigational Site, Plantation, Florida
  - ImClone Investigational Site, Port Saint Lucie, Florida
  - ImClone Investigational Site, St. Petersburg, Florida
  - ImClone Investigational Site, Tampa, Florida
  - ImClone Investigational Site, Albany, Georgia
  - ImClone Investigational Site, Lawrenceville, Georgia
  - ImClone Investigational Site, Park Ridge, Illinois
  - ImClone Investigational Site, Columbia, Maryland
  - ImClone Investigational Site, Rockville, Maryland
  - ImClone Investigational Site, Dearborn, Michigan
  - ImClone Investigational Site, Minneapolis, Minnesota
  - ImClone Investigational Site, Saint Joseph, Missouri
  - ImClone Investigational Site, St Louis, Missouri
  - ImClone Investigational Site, Henderson, Nevada
  - ImClone Investigational Site, Morristown, New Jersey
  - ImClone Investigational Site, Johnson City, New York
  - ImClone Investigational Site, Lake Success, New York
  - ImClone Investigational Site, The Bronx, New York
  - ImClone Investigational Site, Burlington, North Carolina
  - ImClone Investigational Site, Chapel Hill, North Carolina
  - ImClone Investigational Site, Dayton, Ohio
  - ImClone Investigational Site, Middletown, Ohio
  - ImClone Investigational Site, Toledo, Ohio
  - ImClone Investigational Site, Portland, Oregon
  - ImClone Investigational Site, Pittsburgh, Pennsylvania
  - ImClone Investigational Site, Charleston, South Carolina
  - ImClone Investigational Site, Greenville, South Carolina
  - ImClone Investigational Site, Chattanooga, Tennessee
  - ImClone Investigational Site, Nashville, Tennessee
  - ImClone Investigational Site, Arlington, Texas
  - ImClone Investigational Site, Bedford, Texas
  - ImClone Investigational Site, Dallas, Texas
  - ImClone Investigational Site, Fort Worth, Texas
  - ImClone Investigational Site, Houston, Texas
  - ImClone Investigational Site, Plano, Texas
  - ImClone Investigational Site, San Antonio, Texas
  - ImClone Investigational Site, The Woodlands, Texas
  - ImClone Investigational Site, Tyler, Texas
  - ImClone Investigational Site, Rutland, Vermont
  - ImClone Investigational Site, Fairfax, Virginia
  - ImClone Investigational Site, Norfolk, Virginia
  - ImClone Investigational Site, Richmond, Virginia
  - ImClone Investigational Site, Salem, Virginia
  - ImClone Investigational Site, Vancouver, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participant Flow reports participants who discontinued from the study. Participants who died due to any cause and participants who were alive at conclusion of the study but off treatment were considered to have completed the study.
Groups:
- Ramucirumab and Eribulin: Ramucirumab (IMC-1121B) 10 milligrams/kilogram (mg/kg) administered by intravenous (IV) infusion on Day 1 of each 3-week cycle
  Eribulin 1.4 milligrams/square meter (mg/m²) administered by IV bolus on Day 1 and Day 8 of each 3-week cycle
Period: Overall Study
Arm/Group | Ramucirumab and Eribulin | Eribulin Monotherapy
Started | 71 | 70
Received at Least 1 Dose of Study Drug | 69 | 65
Completed | 63 | 57
Not Completed | 8 | 13
Not completed — Withdrawal by Subject | 5 | 8
Not completed — Lost to Follow-up | 1 | 5
Not completed — Other | 1 | 0
Not completed — Investigator's Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Ramucirumab and Eribulin: Ramucirumab (IMC-1121B) 10 mg/kg administered by intravenous (IV) infusion on Day 1 of each 3-week cycle
  Eribulin 1.4 mg/m² administered by IV bolus on Day 1 and Day 8 of each 3-week cycle
- Total: Total of all reporting groups
Arm/Group | Ramucirumab and Eribulin | Eribulin Monotherapy | Total
Number analyzed (Participants) | 71 | 70 | 141
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 62 | 53 | 115
  >=65 years | 9 | 17 | 26
Gender [Count of Participants; unit: Participants]
  Female | 71 | 70 | 141
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 8
  Not Hispanic or Latino | 65 | 67 | 132
  Unknown or Not Reported | 1 | 0 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 1 | 2
  Black or African American | 11 | 8 | 19
  White | 54 | 58 | 112
  Other | 5 | 2 | 7
Region of Enrollment [Number; unit: participants]
  United States | 71 | 70 | 141

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as time from date of randomization until the date of objectively determined progression defined by Response Evaluation Criteria in Solid Tumors (RECIST v1.1) criteria or death from any cause, whichever is first. Progressive disease (PD) defined as ≥20% increase in sum of diameter (SOD) of target lesion with the sum demonstrating an increase of ≥5 mm; appearance of ≥1 new lesions or unequivocal progression of non-target lesions. Participants with no baseline disease assessment were censored at randomization date, regardless of whether or not objectively determined PD or death was observed; participants not known to have died or to have objective progression as of data inclusion cutoff date were censored at last post baseline radiological assessment date or randomization date, if there was no post baseline radiological assessment.
Time Frame: Start of treatment until documented disease progression or death from any cause up to 16.5 months
Population: Intent-to-treat Population (ITT): all participants according to their randomized treatment group. Participants censored: Ramucirumab+Eribulin=14; Eribulin=17.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ramucirumab and Eribulin | Eribulin Monotherapy
Number analyzed (Participants) | 71 | 70
months | 4.4 [3.1 to 6.7] | 4.1 [3.2 to 5.6]

2. Secondary Outcome: Overall Survival (OS) Randomization to Date of Death From Any Cause
Description: Time from the date of randomization to the date of death from any cause. For participants who were not known to have died as of the data-inclusion cut-off date, OS data were censored on the last date the participants were known to be alive prior to that cut-off date.
Time Frame: Randomization to date of death from any cause up to 28.6 months
Population: ITT Population: All randomized participants. Participants censored: Ramucirumab and Eribulin=24 , Eribulin Monotherapy=28
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ramucirumab and Eribulin | Eribulin Monotherapy
Number analyzed (Participants) | 71 | 70
Months | 13.5 [10.4 to 17.9] | 11.5 [9.0 to 17.3]

3. Secondary Outcome: Objective Response Rate (ORR) Percentage of Participants With Measurable Disease Achieving a Best Overall Response of Partial Response (PR) or Complete Response (CR)
Description: ORR was defined as the percentage of participants with measurable disease achieving a best overall response of PR or CR as defined by RECIST v.1.1. CR defined as disappearance of all lesions and pathological lymph nodes reduction in short axis to <10 mm. PR was defined as ≥30% decrease in SOD of target lesions. Participants who did not have any post baseline tumor response assessments for any reason were considered non-responders and included in the denominator when calculating the response rate. ORR for each treatment arm calculated as: [(CR + PR in the treatment arm) divided by (total number of participants in the treatment arm)] x 100.
Time Frame: Start of treatment until documented CR or PR up to 16.5 months
Population: ITT population: all participants according to their randomized treatment group.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ramucirumab and Eribulin | Eribulin Monotherapy
Number analyzed (Participants) | 71 | 70
percentage of participants | 19.7 [11.2 to 30.9] | 24.3 [14.8 to 36.0]

4. Secondary Outcome: Duration of Response (DOR) Time of Response to Progressive Disease
Description: DOR was measured from the time criteria were met for first objectively recorded CR or PR until first date criteria for PD was met or death. Response defined using RECIST v1.1 criteria. CR defined as disappearance of all lesions and pathological lymph nodes reduction in short axis to <10 mm. PR was defined as ≥30% decrease in sum of diameter (SOD) of target lesions. PD defined ≥20% increase in SOD of target lesion with the sum demonstrating an increase of ≥5 mm; appearance of ≥1 new lesions or unequivocal progression of non-target lesions. Participants who were not known to have died and who did not have PD were censored at the date of the last tumor assessment prior to the date of any subsequent systemic anticancer therapy.
Time Frame: Time from Observed CR or PR to PD up to 12.1 months
Population: ITT population: all participants according to their randomized treatment group and who had CR or PR. Participants censored: Ramucirumab+Eribulin=1, Eribulin=3.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ramucirumab and Eribulin | Eribulin Monotherapy
Number analyzed (Participants) | 14 | 17
months | 5.5 [3.1 to 7.1] | 3.0 [1.4 to 4.4]

5. Secondary Outcome: Change in Tumor Size (CTS)
Description: CTS was defines as the change from baseline measurement of target lesions to the post treatment measurement in participants with measurable disease. Change was assessed using radiographic imagining. Log ratio calculated as: log of (tumor size post baseline) divided by (tumor size at baseline). A negative result indicated a shrinking tumor.
Time Frame: Baseline, 6 weeks
Population: All participants with measurable disease at baseline and at 6 weeks.
Measure: Mean (Standard Deviation); unit: log ratio
Arm/Group | Ramucirumab and Eribulin | Eribulin Monotherapy
Number analyzed (Participants) | 43 | 39
log ratio | -0.20 (0.33) | -0.20 (0.28)

6. Secondary Outcome: Number of Participants With Anti-Ramucirumab Antibodies
Description: The number of participants who developed treatment-emergent antibody responses after baseline. The antibody test can produce positive results in participants without ramucirumab exposure. Treatment emergent anti-ramucirumab antibody positive was defined as: when baseline titer was greater than 0 and post baseline titer was equal to or greater than 4-fold the baseline titer or if the baseline titer was not detected and post baseline titer is equal to or greater than a value of 20.
Time Frame: Day 1 of Cycle 1, Cycle 3, Cycle 5 and 30 days after last dose of study drug up to 17.7 months
Population: All randomized participants who received at least 1 dose of study drug and assessed for treatment emergent antibodies.
Measure: Number; unit: participants
Arm/Group | Ramucirumab and Eribulin | Eribulin Monotherapy
Number analyzed (Participants) | 61 | 41
participants | 4 | 2

7. Other Pre Specified Outcome: Number of Participants With Adverse Events (AE) and Participants Who Died
Description: Participants who died or who had clinically significant events defined as serious AEs (SAEs) and other non-serious AEs (regardless of causality). A summary of SAEs and other non-serious AEs, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Baseline up to end of treatment and within 30 days of last dose of study drug (22.6 months)
Population: All randomized participants who received at least 1 dose of study drug and according to the treatment received.
Measure: Number; unit: participants
Arm/Group | Ramucirumab and Eribulin | Eribulin Monotherapy
Number analyzed (Participants) | 69 | 65
participants
  SAE | 26 | 12
  Other non-SAE | 68 | 65
  Died | 30 | 32

ADVERSE EVENTS:
Description: SAE's and other non-SAE's are treatment emergent.
Arm/Group | Ramucirumab and Eribulin | Eribulin Monotherapy
Serious Adverse Events (participants affected / at risk) | 26/69 | 12/65
Other Adverse Events (participants affected / at risk) | 67/69 | 64/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ramucirumab and Eribulin (N=69) | Eribulin Monotherapy (N=65)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 4 (4) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 2 (2)
Ascites (Gastrointestinal disorders) | 2 (2) | 2 (2)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 2 (3) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Drug withdrawal syndrome (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Oedema (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pleural infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Systemic candida (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ramucirumab and Eribulin (N=69) | Eribulin Monotherapy (N=65)
Anaemia (Blood and lymphatic system disorders) | 13 (20) | 16 (37)
Leukopenia (Blood and lymphatic system disorders) | 4 (15) | 8 (31)
Neutropenia (Blood and lymphatic system disorders) | 27 (71) | 29 (75)
Thrombocytopenia (Blood and lymphatic system disorders) | 8 (17) | 4 (13)
Abdominal distension (Gastrointestinal disorders) | 4 (6) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 9 (17) | 9 (9)
Abdominal pain upper (Gastrointestinal disorders) | 4 (5) | 0 (0)
Ascites (Gastrointestinal disorders) | 4 (5) | 0 (0)
Constipation (Gastrointestinal disorders) | 20 (25) | 19 (21)
Diarrhoea (Gastrointestinal disorders) | 17 (21) | 10 (19)
Dyspepsia (Gastrointestinal disorders) | 5 (7) | 6 (7)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 (4) | 4 (4)
Nausea (Gastrointestinal disorders) | 28 (48) | 27 (41)
Stomatitis (Gastrointestinal disorders) | 8 (11) | 4 (7)
Vomiting (Gastrointestinal disorders) | 19 (32) | 17 (24)
Asthenia (General disorders) | 4 (6) | 2 (4)
Fatigue (General disorders) | 43 (77) | 38 (53)
Local swelling (General disorders) | 3 (4) | 4 (5)
Mucosal inflammation (General disorders) | 6 (7) | 3 (3)
Oedema peripheral (General disorders) | 10 (13) | 11 (12)
Pain (General disorders) | 5 (6) | 4 (4)
Pyrexia (General disorders) | 14 (21) | 5 (9)
Seasonal allergy (Immune system disorders) | 4 (4) | 2 (2)
Sinusitis (Infections and infestations) | 7 (10) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 6 (6) | 9 (9)
Urinary tract infection (Infections and infestations) | 2 (2) | 7 (7)
Alanine aminotransferase increased (Investigations) | 10 (11) | 5 (6)
Aspartate aminotransferase increased (Investigations) | 10 (12) | 6 (9)
Blood alkaline phosphatase increased (Investigations) | 4 (4) | 5 (7)
Neutrophil count decreased (Investigations) | 5 (19) | 8 (27)
Weight decreased (Investigations) | 4 (4) | 2 (3)
White blood cell count decreased (Investigations) | 6 (17) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 19 (20) | 12 (13)
Dehydration (Metabolism and nutrition disorders) | 10 (15) | 7 (8)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (12) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 6 (9) | 7 (8)
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 (6) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 8 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (9) | 4 (12)
Bone pain (Musculoskeletal and connective tissue disorders) | 7 (9) | 4 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 (6) | 3 (4)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 4 (7)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (8) | 5 (10)
Dizziness (Nervous system disorders) | 8 (10) | 7 (8)
Dysgeusia (Nervous system disorders) | 6 (6) | 4 (5)
Headache (Nervous system disorders) | 27 (39) | 10 (16)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 4 (4)
Peripheral motor neuropathy (Nervous system disorders) | 2 (3) | 5 (8)
Peripheral sensory neuropathy (Nervous system disorders) | 15 (23) | 17 (30)
Anxiety (Psychiatric disorders) | 4 (7) | 3 (3)
Depression (Psychiatric disorders) | 3 (4) | 6 (7)
Insomnia (Psychiatric disorders) | 9 (9) | 6 (6)
Proteinuria (Renal and urinary disorders) | 4 (4) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 12 (15)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 (18) | 14 (21)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (5)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 20 (22) | 15 (16)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (5)
Rash (Skin and subcutaneous tissue disorders) | 5 (10) | 3 (4)
Flushing (Vascular disorders) | 4 (4) | 1 (1)
Hypertension (Vascular disorders) | 9 (10) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators agreed to delay independently publishing or disclosing data, findings or conclusions from the study except as part of a multi-center publication. Upon study publication or if the draft publication is not produced within approximately 6 months of the final report of the study results, investigators may independently publish, subject to confidential information review/redaction by sponsor. The sponsor may request publication delay up to 90 days to seek patent protection.